CLINICAL TRIAL: NCT02564978
Title: Evaluation of Oral Minocycline in the Treatment of Geographic Atrophy Associated With Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150202; 15-EI-0202
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2022-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: Eye Disease; Degenerative
MeSH Terms: conditions — Macular Degeneration; Eye Diseases | interventions — Minocycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Minocycline (Experimental): Oral administration of minocycline.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Adult participants will be instructed to take their prescribed IP orally two times a day, once in the morning and once in the evening, approximately 12 hours apart. The capsules will be dispensed to the participant in a tight, light-resistant container as defined in the USP in three-month supply aliquots. Starting at Month 9 and continuing at Month 12, a three-month supply will be dispensed to the participant during the study visit or mailed to the participant. Participants will be given an instruction sheet for taking the prescribed IP. Starting at Month 15 participants will receive two bottles for a six-month supply. The IP should be stored between 15-30 degrees C (or 59-86 degrees F).They should be protected from light, moisture, and excessive heat. Participants will be required to bring their bottles of IP to each appropriate visit for capsule counts for compliance monitoring.

SUMMARY:
Background:

Age-related macular degeneration (AMD) is the main reason older people lose their vision. It affects the macula, the center of the retina needed for sharp, clear vision. Researchers want to see if an antibiotic can help people with an advanced form of AMD, Geographic Atrophy (GA).

Objective:

To see if minocycline is safe for people with GA and if it helps preserve their vision.

Eligibility:

People age 55 and older who have GA in at least one eye.

Design:

Participants will be screened with physical exam, medical history, blood tests, and eye exam.

Participants will take minocycline. They will take 1 pill twice a day for at least 3 years.

Participants will have a minimum of 11 study visits. (But they are not every 3 months.). At each visit, participants will have a medical history. They may have:

Blood tests.

Eye exam. Vision, eye pressure, and eye movements will be checked. The pupils may be dilated. The inside of the eyes may be photographed.

Their thyroid gland felt while they swallow.

Microperimetry. They will sit in front of a computer and press a button when they see a light on the screen.

Fluorescein angiography. An intravenous line (IV) will be placed in an arm vein. A dye called fluorescein will be placed in the IV and travel through the veins to the blood vessels in the eyes. A camera will take pictures of the dye as it flows through the eye blood vessels.

DETAILED DESCRIPTION:
Objective: Age-related macular degeneration (AMD), the leading cause of blindness in people over age 65 in the United States, is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment of central visual acuity (VA). AMD occurs in two general forms, one of which involves choroidal neovascularization (CNV) with subsequent formation of a disciform scar. This is often referred to as the neovascular or wet form. A second form, the subject of this study, is termed dry /atrophic macular degeneration or otherwise geographic atrophy (GA) and involves a slow progressive atrophy of retinal pigment epithelial (RPE) cells and photoreceptors in the macula, also resulting in central vision loss. GA is estimated to affect up to one million persons in the U.S. and there is no current treatment that can prevent its onset or retard its progression.

While the etiology of GA is not completely understood, inflammatory processes involving the activation of resident immune cells of the retina called microglia is likely to contribute. Minocycline inhibits the activation of microglia which produce inflammatory factors implicated in GA development. The objective of this study is to investigate the safety and possible efficacy of oral minocycline in patients with GA.

Study Population: Forty-five participants with unilateral or bilateral GA associated with AMD will be enrolled. However, up to an additional 15 participants may be enrolled to replace participants who may withdraw from the study prior to reaching the Month 33 visit.

Design: This is a multi-center, prospective, single-arm, Phase II study to evaluate minocycline as a potential treatment to decrease the rate of worsening of GA associated with AMD.

Participants will undergo a nine-month run-in phase prior to receiving investigational product (IP). During this run-in phase, participants will have a total of four pre-treatment visits. Following the run-in phase, beginning at Month 9, participants will receive an oral dose of 100 mg of minocycline twice daily for 36 months. There will be a common termination date, which will take place when the last recruited participant has received 36 months of treatment. Participants who were recruited in the earlier part of the study will continue treatment and be followed every six months until the common termination date. However, participants may complete participation in the study as early as Month 45, at the discretion of the investigator.

Outcome Measures: The primary outcome is the rate of change in area of GA based on grading by an external Reading Center of fundus autofluorescence (FAF) images in the assigned study eye. The primary outcome will compare the rates of GA area expansion as determined on FAF images before and following the initiation of IP until 24 months of treatment. Secondary outcomes will compare differences in rates of change in best-corrected visual acuity (BCVA), low-luminance VA, area of GA based on FAF (using a different statistical approach compared to primary outcome) and fundus photography. The exploratory outcome will compare the difference in the rate of change in macular sensitivity as measured using microperimetry. This outcome was originally a secondary outcome when the clinical trial participants were enrolled, since these represent visual function data corresponding closely to areas affected by geographic atrophy. Hence, changes in microperimetry data over time might be well placed to support changes in structural data over time, as geographic atrophy lesions undergo enlargement. In the original Statistical Analysis Plan, the intention was that "Macular sensitivity, as measured on microperimetry, will be evaluated in a similar manner as BCVA", (i.e., Mean rate of change in BCVA during the treatment phase will be compared to the mean rate of change in BCVA during the run-in phase using Student s paired t-test ). However, microperimetry data (represented by multiple numerical values, one for each anatomical location, at each time-point) are much more complex than BCVA data (represented by a single numerical value at each time-point). The originally proposed statistical treatment is therefore not suitable. In addition, the study team is not aware of any established methods accepted by the community for analyzing microperimetry data, unlike the situation for BCVA. Indeed, the microperimetry acquisition pattern used in GA MIN is unique and was developed specifically for this trial. It therefore needs its own dedicated set of statistical analyses (which may need several iterations), rather than pre-specified and widely accepted analyses that could be detailed in advance in the Statistical Analysis Plan. For these reasons, although the original intention was for the microperimetry data to represent a secondary outcome measure, it is better suited to an exploratory outcome measure. Safety outcomes will include the number and severity of adverse events (AEs). Ocular safety outcomes will be indicated by changes in VA, ocular surface changes, intraocular inflammation and any other ocular changes not consistent with the natural progression of GA.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable:

* Participant must be 55 years of age or older.
* Participant must understand and sign the protocol s informed consent document.
* Participant must have evidence of early or intermediate AMD as defined by characteristic presence of drusen and/or pigmentary changes.
* Participant must be able to swallow capsules.
* Participant must have normal renal function and liver function or have mild abnormalities not above grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
* Participant must agree to minimize exposure to sunlight or artificial ultraviolet (UV) rays and to wear protective clothing, sunglasses and sunscreen (minimum sun protection factor (SPF) 15) if s/he must be out in the sun.
* Any female participant of childbearing potential (see Appendix 1 for definition) must have a negative pregnancy test at screening and be willing to undergo pregnancy tests throughout the study.
* Any female participant of childbearing potential (see Appendix 1 for definition) and any male participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent* from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for at least one week after investigational product (IP) discontinuation. Acceptable methods of contraception include:

  1. hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
  2. intrauterine device,
  3. barrier methods (diaphragm, condom) with spermicide, or,
  4. surgical sterilization (hysterectomy or tubal ligation).

     * Abstinence is only acceptable when it is the participant s preferred and usual lifestyle choice. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

* Participant is actively receiving study therapy in another investigational study.
* Any female participant of childbearing potential (see Appendix 1 for definition) that is pregnant, breast-feeding or planning to become pregnant during the study.
* Participant is expected to be unable to comply with study procedures or follow-up visits.
* Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve (e.g., ethambutol, chloroquine, or hydroxychloroquine).
* Participant has a condition that would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control) by interfering with the participant s ability to engage in the required protocol evaluation and testing and/or comply with study visits.
* Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
* Participant has a history of chronic hepatitis or liver failure.
* Participant has a history of thyroid cancer.
* Participant has an allergy or hypersensitivity to minocycline or any drug in the tetracycline family.
* Participant is currently taking minocycline or another tetracycline medication.
* Participant is taking any medication that could adversely interact with minocycline such as methoxyflurane.
* Participant has a prior history of idiopathic intracranial hypertension.

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

* The study eye must have greater than 1/2 disc area (approximately 1 mm(2)) of GA compatible with dry AMD. GA is defined as one or more well-defined and often circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial depigmentation may be classified as early GA. The GA in the study eye must be able to be photographed in their entirety, and it must not be contiguous with any areas of peripapillary atrophy, which can complicate area measurements.
* The total area of GA lesions combined should be less than 7.0 MPS disc areas (DA) (17.78 mm(2)) as evident on FAF imaging.
* The VA of the study eye should be greater than or equal to19 E-ETDRS letters (i.e., 20/400 or better).
* The study eye must have clarity of ocular media and degree of pupil dilation sufficient to permit adequate fundus photographs.

STUDY EYE EXCLUSION CRITERIA:

* Current evidence of choroidal neovascularization (CNV) as determined by the treating physician or a history of treatments for CNV
* Evidence of retinal atrophy due to causes other than atrophic AMD.
* Current evidence or history of ocular disorders in the study eye that in the opinion of the investigator confounds study outcome measures, including (but not limited to):

  1. non-proliferative diabetic retinopathy involving 10 or more hemorrhages or microaneurysms, or active proliferative diabetic retinopathy
  2. Branch or central retinal vein or artery occlusion
  3. Macular hole
  4. Pathologic myopia
  5. Uveitis
  6. Pseudovitelliform maculopathy
* History of vitreoretinal surgery.
* Need for ocular surgery during the course of the study.
* Recent history of lens removal (less than 3 months) or Yttrium Aluminum Garnet (YAG) laser capsulotomy (less than 1 month).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiarnan DL Keenan, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mukherjee S, Vance E, von der Emde L, Arunachalam T, De Silva T, Thavikulwat AT, Orndahl C, Nyaiburi C, Abraham M, Hammel K, Sadda SR, Chew EY, Pfau M, Wong WT, Jeffrey BG, Keenan TDL. Variation in Mesopic Retinal Sensitivity Relative to Distance from Geographic Atrophy in Age-Related Macular Degeneration. Ophthalmol Sci. 2025 Jul 8;5(6):100879. doi: 10.1016/j.xops.2025.100879. eCollection 2025 Nov-Dec. PMID 40837068
- [Result] Keenan TDL, Bailey C, Abraham M, Orndahl C, Menezes S, Bellur S, Arunachalam T, Kangale-Whitney C, Srinivas S, Karamat A, Nittala M, Cunningham D, Jeffrey BG, Wiley HE, Thavikulwat AT, Sadda S, Cukras CA, Chew EY, Wong WT. Phase 2 Trial Evaluating Minocycline for Geographic Atrophy in Age-Related Macular Degeneration: A Nonrandomized Controlled Trial. JAMA Ophthalmol. 2024 Apr 1;142(4):345-355. doi: 10.1001/jamaophthalmol.2024.0118. PMID 38483382
- [Result] Mukherjee S, Arunachalam T, Duic C, Abraham M, Orndahl C, Menezes S, Agron E, Pfau M, de Silva T, Bailey C, Thavikulwat AT, Bellur S, Sadda SR, Chew EY, Jeffrey BG, Wong WT, Keenan TDL. Structure-Function Relationships in Geographic Atrophy Based on Mesopic Microperimetry, Fundus Autofluorescence, and Optical Coherence Tomography. Transl Vis Sci Technol. 2025 Feb 3;14(2):7. doi: 10.1167/tvst.14.2.7. PMID 39908134
- [Result] Arunachalam T, Abraham M, Orndahl C, Menezes S, Mukherjee S, Duic C, Prasad M, Siddig F, Bellur S, Thavikulwat AT, Bailey C, Sadda SR, Wong WT, Chew EY, Jeffrey BG, Keenan TDL. Longitudinal Analysis of Mesopic Microperimetry in a Phase II Trial Evaluating Minocycline for Geographic Atrophy. Ophthalmol Sci. 2025 Apr 1;5(5):100783. doi: 10.1016/j.xops.2025.100783. eCollection 2025 Sep-Oct. PMID 40417242
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-EI-0202.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to forty-five (45) participants with unilateral or bilateral geographic atrophy (GA) associated with age-related macular degeneration (AMD) will be enrolled. Up to an additional 15 participants may be enrolled to replace participants who withdraw from the study prior to reaching the Month 33 visit. Participants with GA in at least one eye that is associated with AMD were enrolled. Enrollment closed at the National Eye Institute and Bristol Eye Hospital on December 31, 2019.
Pre-assignment Details: Participants must have at least one eye meeting all inclusion criteria and none of the exclusion criteria as defined in the protocol. For participants with two qualifying eyes, the fellow (non-study) eye will be noted as a "qualifying fellow eye." All eligible participants undergo treatment starting at Month 9 (e.g., are a part of the "Minocycline" group). The IP used in the study is oral minocycline and is not anticipated to differentially treat participant eyes.
Groups:
- Minocycline: Oral administration of minocycline.
  Minocycline: Participants underwent a nine-month run-in phase without taking minocycline. At Month 9, they were instructed to begin taking 100 mg of oral minocycline twice daily until study termination, after a minimum of 36 months on IP. Starting at Month 9 and continuing at Month 12, a three-month supply was dispensed to the participant during the study visit or mailed to the participant. Starting at Month 15 participants received two bottles for a six-month supply. Participants were required to bring their bottles of IP to each appropriate visit for capsule counts for compliance monitoring. Participants could complete participation in the study and discontinue treatment as early as Month 45 (36 months of treatment phase). At the conclusion of the study, participants were no longer eligible to receive IP under this protocol.
Period: Overall Study
Arm/Group | Minocycline
Started | 37
Completed Run-in Phase (Completed Run-in Phase and Initiated Treatment Phase) | 36
Completed Month 33 Visit (Primary outcome is assessed at Month 33.) | 21
Completed Month 45 Visit (Minimum required follow-up is through Month 45. Common termination date is reached when the last enrolled participant completes the study through Month 45. Prior to Amendment L, follow-up beyond Month 45 may be completed for those participants enrolled at the beginning of the study and continue on study until the common termination date. As of Amendment L, participants could complete the study per-protocol prior to the common termination date and as early as Month 45 at the discretion of the PI.) | 10
Completed Month 57 Visit (Minimum required follow-up is through Month 45. Common termination date is reached when the last enrolled participant completes the study through Month 45. Prior to Amendment L, follow-up beyond Month 45 may be completed for those participants enrolled at the beginning of the study and continue on study until the common termination date. As of Amendment L, participants could complete the study per-protocol prior to the common termination date and as early as Month 45 at the discretion of the PI.) | 4
Completed | 5
Not Completed | 32
Not completed — Adverse Event | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 15
Not completed — Early Study Closure | 2
Not completed — Other Reason | 5

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
  Europe | 7
Square Root of Total Area of Definite Decreased Autofluorescence [Mean (Standard Deviation); unit: mm] — Baseline measurement of square-root of total area definite decreased autofluorescence in the study eye as assessed by fundus autofluorescence. Population: For one participant, GA area could not be graded at baseline due to poor image quality.
  mm
    number analyzed (Participants) | 36
    (all) | 2.5 (0.9)
Square Root of Total Area of Macular GA [Mean (Standard Deviation); unit: mm] — Baseline measurement of square-root of total area macular GA in the study eye as assessed by color fundus photography. Population: Summary based on participants who received at least one dose of the study drug. Due to a software issue, some CFP images could not be graded for quantitative measures.
  mm
    number analyzed (Participants) | 31
    (all) | 2.5 (1.0)
Best-Corrected Visual Acuity Total Letters Read [Mean (Standard Deviation); unit: letters read] — Baseline measurement of BCVA total letters read in the study eye. Population: Summary based on participants who received at least one dose of the study drug.
  letters read
    number analyzed (Participants) | 35
    (all) | 64.4 (14.3)
Low Luminance Visual Acuity Total Letters Read [Mean (Standard Deviation); unit: letters read] — Baseline measurement of LLVA total letters read in the study eye. Population: Summary based on participants who received at least one dose of the study drug.
  letters read
    number analyzed (Participants) | 35
    (all) | 51.5 (16.0)
Central Retinal Thickness [Mean (Standard Deviation); unit: um] — Baseline measurement of central retinal thickness in the study eye as assessed by Optical Coherence Tomography. Population: Summary based on participants who received at least one dose of the study drug.
  um
    number analyzed (Participants) | 34
    (all) | 123.1 (67.5)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Square-Root Transformed GA Area Expansion Rates in the Study Eye Between the Treatment Phase and Run-in Phase Based on Fundus Autofluorescence (FAF)
Description: The difference in the square-root transformed GA area expansion rates in the study eye based on fundus autofluorescence (FAF) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) was compared using a linear spline regression model with a fixed knot at Month 9, at a Type I error rate of 2.5%.
Time Frame: Run-in phase (baseline to Month 9) before initiation of IP and 24 months treatment phase after initiation of IP (Month 9 to Month 33)
Population: Participants in the enrolled population (all participants enrolled in the study, regardless of compliance, follow-up or treatment received) with at least one data point for the study eye.
Measure: Least Squares Mean (Standard Error); unit: mm/year
Units Other Than Participants: Eyes
Groups:
- Minocycline: Participants, ages 55 years and older, with unilateral or bilateral Geographic Atrophy (GA) associated with atrophic Age-Related Macular Degeneration (AMD) underwent a nine-month run-in period prior to receiving IP. Starting at Month 9 (IP start visit), participants received 100 mg minocycline orally twice a day for a total of at least 36 months (i.e., through Month 45).
Arm/Group | Minocycline
Number analyzed (Participants) | 36
Number analyzed (Eyes) | 36
mm/year | -0.03 (0.03)
Statistical Analysis 1: Comparison: Minocycline; Analysis: linear spline regression with fixed knot @ Month 9 on study eyes alone. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between treatment phase & run-in phase >= 0. Square root transformation used to satisfy the linear trend assumption. Missing values: treated as missing completely at random. Covariance structure of random effect that provided best model fit chosen (Spatial Power). One-sided Type I error rate: 2.5%; Test type: Superiority; p = 0.39, Mixed Models Analysis — Result of statistical analyses were considered significant if the p-value from the one-sided test was <0.025. No adjustments for multiplicity were made; Slope = -0.03, Standard Error of Mean 0.03 — The estimate was the difference in rates of change in mean of appropriately transformed GA area between the treatment phase and run-in phase

2. Secondary Outcome: Difference in Square-root Transformed GA Area Expansion Rates Between the Treatment Phase and Run-in Phase Based on Fundus Autofluorescence (FAF)
Description: The difference in the square-root transformed of GA area expansion rates based on fundus autofluorescence (FAF) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) in the study eyes alone, the qualifying fellow eyes alone, and the study eyes and qualifying fellow eyes together, analyzed via a two-sided Student's paired t-test at a Type I error rate of 5%.
Time Frame: as for outcome 1
Population: Participants in the enrolled population (all participants enrolled in the study, regardless of compliance, follow-up or treatment received) with data for the respective eyes at Baseline, Month 9 and Month 33 for the respective analysis.
Measure: Mean (95% Confidence Interval); unit: mm/year
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 33
mm/year
  Study eye: number analyzed (Eyes) | 21
  Study eye | -0.01 [-0.06 to 0.03]
  Qualifying fellow eye: number analyzed (Participants) | 12
  Qualifying fellow eye: number analyzed (Eyes) | 12
  Qualifying fellow eye | -0.1 [-0.24 to 0.04]
  Avg. of Study eye and Qualifying fellow eye | -0.04 [-0.09 to 0.01]
Statistical Analysis 1: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study eyes alone. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.48, t-test, 2 sided — Result of statistical analyses were considered significant if the p-value from the two-sided Student's paired t-test was <0.05. No adjustments for multiplicity were made; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.03]
Statistical Analysis 2: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on qualifying fellow eyes alone. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.15, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.24 to 0.04]
Statistical Analysis 3: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study and qualifying fellow eyes (Study eye + QFE) together. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.15, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.09 to 0.01] — No. of units analyzed = no. of study eyes + no. qualifying fellow eyes (QFE). However, the value contributing to analysis is the avg. of study eye & QFE from a participant if both values are available, otherwise equal to eye with data available

3. Secondary Outcome: Difference in the Square-root Transformed GA Area Expansion Rates Between the Treatment Phase and Run-in Phase Based on Color Fundus Photography (CFP)
Description: The difference in the square-root transformed of GA area expansion rates based on color fundus photography (CFP) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) in the study eyes alone, qualifying fellow eyes alone, and study eyes and qualifying fellow eyes together was compared using a linear spline regression model with a fixed knot at Month 9 at a Type I error rate of 2.5%.
Time Frame: as for outcome 1
Population: Participants in the Per-protocol population 2 (Participants who completed at least three follow-up visits during the 24-month treatment phase and did not discontinue treatment prior to the completion of at least three follow-up visits) with data for the respective eyes, for the respective analysis.
Measure: Least Squares Mean (Standard Error); unit: mm/year
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 26
Number analyzed (Eyes) | 41
mm/year
  Study eye: number analyzed (Eyes) | 26
  Study eye | 0.03 (0.05)
  Qualifying fellow eye: number analyzed (Participants) | 15
  Qualifying fellow eye: number analyzed (Eyes) | 15
  Qualifying fellow eye | -0.06 (0.08)
  Study eye + Qualifying fellow eye | -0.01 (0.04)
Statistical Analysis 1: Comparison: Minocycline; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.61, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 0.03, Standard Error of Mean 0.05 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Minocycline; Analysis: linear spline regression with fixed knot @ Month 9 on qualifying fellow eyes alone. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between treatment phase & run-in phase >= 0. Square root transformation used to satisfy the linear trend assumption. Missing values: treated as missing completely at random. Covariance structure of random effect that provided best model fit chosen (Spatial Power). One-sided Type I error rate: 2.5%; Test type: Superiority; p = 0.43, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = -0.06, Standard Error of Mean 0.08 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Minocycline; Analysis: linear spline regression with fixed knot @ Month 9 on study and qualifying fellow eyes together. Null hypothesis: difference in rates of change in mean of square-root transformed GA area between treatment phase & run-in phase >= 0. Square root transformation used to satisfy the linear trend assumption. Missing values: treated as missing completely at random. Covariance structure of random effect that provided best model fit chosen (Spatial Power). One-sided Type I error rate: 2.5%; Test type: Superiority; p = 0.89, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = -0.01, Standard Error of Mean 0.04 — Study eye + QFE: study & qualifying fellow eyes analyzed as separate observations. Estimate: difference in rate of change in mean of appropriately transformed GA area between treatment and run-in phase

4. Secondary Outcome: Difference in the Mean Rate of Change in Best Corrected Visual Acuity (BCVA) Between the Treatment Phase and Run-in Phase
Description: The difference in the mean rate of change in Best Corrected Visual Acuity (BCVA) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) for the study eyes alone, the qualifying fellow eyes alone, and the study eyes and qualifying fellow eyes together, analyzed via a two-sided Student's paired t-test at a Type I error rate of 5%.
Time Frame: as for outcome 1
Population: Participants in the Per-protocol population 2 (Participants who completed at least three follow-up visits during the 24-month treatment phase and did not discontinue treatment prior to the completion of at least three follow-up visits) with data for the respective eyes at Baseline, Month 9 and Month 33 for the respective analysis.
Measure: Mean (95% Confidence Interval); unit: letters read/month
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 27
letters read/month
  Study eye: number analyzed (Eyes) | 18
  Study eye | 0.2 [-0.4 to 0.9]
  Qualifying fellow eye: number analyzed (Participants) | 9
  Qualifying fellow eye: number analyzed (Eyes) | 9
  Qualifying fellow eye | -0.3 [-0.8 to 0.2]
  Avg. of Study eye and Qualifying fellow eye | 0.2 [-0.4 to 0.8]
Statistical Analysis 1: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study eyes alone. Null hypothesis: difference in the mean rates of change in BCVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.44, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9]
Statistical Analysis 2: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on qualifying fellow eyes alone. Null hypothesis: difference in the mean rates of change in BCVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.21, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.2]
Statistical Analysis 3: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study and qualifying fellow eyes together (Study eye + QFE). Null hypothesis: difference in the mean rates of change in BCVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.52, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.8] — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Difference in the Mean Rate of Change in Low-Luminance Visual Acuity (LLVA) Between the Treatment Phase and Run-in Phase
Description: The difference in the mean rate of change in Low-Luminance Visual Acuity (LLVA) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) for the study eyes alone, the qualifying fellow eyes alone, and the study eyes and qualifying fellow eyes together, analyzed via a two-sided Student's paired t-test at a Type I error rate of 5%.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: letters read/month
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 26
letters read/month
  Study eye: number analyzed (Eyes) | 17
  Study eye | 0.2 [-0.4 to 0.9]
  Qualifying fellow eye: number analyzed (Participants) | 9
  Qualifying fellow eye: number analyzed (Eyes) | 9
  Qualifying fellow eye | -0.4 [-0.9 to 0.1]
  Avg. of Study eye and Qualifying fellow eye | 0.2 [-0.4 to 0.7]
Statistical Analysis 1: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study eyes alone. Null hypothesis: difference in the mean rates of change in LLVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9]
Statistical Analysis 2: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on qualifying fellow eyes alone. Null hypothesis: difference in the mean rates of change in LLVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.09, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 3: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study and qualifying fellow eyes together (Study eye + QFE). Null hypothesis: difference in the mean rates of change in LLVA between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.54, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.7] — [estimate comment as in outcome 2, analysis 3]

6. Secondary Outcome: Difference in the Mean Rate of Change of Central Retinal Thickness as Measured on Optical Coherence Tomography (OCT) Between the Treatment Phase and Run-in Phase
Description: The difference in the mean rate of change of central retinal thickness as measured on Optical Coherence Tomography (OCT) between the treatment phase (Month 9 to Month 33) and the run-in phase (baseline to Month 9) for the study eyes alone, the qualifying fellow eyes alone, and the study eyes and qualifying fellow eyes together, analyzed via a two-sided Student's paired t-test at a Type I error rate of 5%.
Time Frame: as for outcome 1
Population: Participants in the Per-protocol population 2 (Participants who completed at least three follow-up visits during the 24-month treatment phase and did not discontinue treatment prior to the completion of at least three follow-up visits) with data for the respective eyes at Baseline, Month 9 and Month 33 for the respective analysis. Participants may have data from the qualifying fellow eye only.
Measure: Mean (95% Confidence Interval); unit: μm/month
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 18
Number analyzed (Eyes) | 26
μm/month
  Study eye: number analyzed (Participants) | 17
  Study eye: number analyzed (Eyes) | 17
  Study eye | 0.7 [-0.4 to 1.8]
  Qualifying fellow eye: number analyzed (Participants) | 9
  Qualifying fellow eye: number analyzed (Eyes) | 9
  Qualifying fellow eye | 1.8 [0.4 to 3.1]
  Avg. of Study eye and Qualifying fellow eye | 1.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study eyes alone. Null hypothesis: difference in the mean rate of change of central retinal thickness as measured on OCT between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.20, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.4 to 1.8]
Statistical Analysis 2: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on qualifying fellow eyes alone. Null hypothesis: difference in the mean rate of change of central retinal thickness as measured on OCT between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority; p = 0.02, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [0.4 to 3.1]
Statistical Analysis 3: Comparison: Minocycline; Analysis: two-sided Student's paired t-test on study and qualifying fellow eyes together (Study eye + QFE). Null hypothesis: difference in the mean rate of change of central retinal thickness as measured on OCT between the treatment phase and run-in phase is not equal to 0. Missing values: treated as missing completely at random. Two-sided Type I error rate: 5%; Test type: Superiority — Number of eyes contributing to this analysis exceeds the number of eyes contributing to the study eye only analysis since one participant had relevant data for the qualifying fellow eye but not the study eye; p = 0.06, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 2.0] — [estimate comment as in outcome 2, analysis 3]

ADVERSE EVENTS:
Time Frame: Participants enrolled at the United States site are assessed for AEs starting at Month 9, after IP initiation, for up to 48 months. Participants enrolled at the European site are assessed for AEs starting at the baseline visit for up to 57 months.
Arm/Group | Minocycline
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 8/37
Other Adverse Events (participants affected / at risk) | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=37)
Tachycardia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (2)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=37)
Blood thyroid stimulating hormone increased (Investigations) | 15 (18)
Blood thyroid stimulating hormone decreased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
SARS-CoV 2 test positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (7)
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Sebaceous glands overactivity (Skin and subcutaneous tissue disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Meibomian gland dysfunction (Eye disorders) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Keratopathy (Eye disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dementia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Potential disadvantages of study design (each participant eye serves as own control): long study period, requirement for participants to wait to begin treatment, and more complex interpretation of safety data. Potential limitations of study: discontinuation of study drug/study in number of participants (accounted for in sample size calculations), absence of assays to analyze microglial activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT02564978/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02564978/SAP_001.pdf
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT02564978/ICF_002.pdf